CLINICAL TRIAL: NCT07083076
Title: Early Introduction of Regular Diet Versus Extended Low Residue Restriction After Colon Surgery
Brief Title: Regular Diet Versus Extended Low Residue After Colon Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Andrea Zimmern, Assistant Professor of Surgery Donald and Barbara Zucker School of Medicine at Hofstra/Northwell, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-0448
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-07

CONDITIONS: Colon Resection
Keywords: postoperative diet; low residue diet; colon resection with anastomosis

STUDY DESIGN:
Intervention Model Description: Group A: 10 day low residue diet resection after colon resection surgery Group B: 6 week low residue diet resection after colon resection surgery
  Groups are stratified by hospital, side of colon resected, and biological sex
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10 day low residue diet restriction after surgery (Experimental): 10 day low residue diet restriction after surgery
  Interventions: Other: Short term (10 day) low residue diet restriction
- 6 week low residue diet restriction after surgery (Other): Usual care arm
  Interventions: Other: 6 week low residue diet restriction

INTERVENTIONS:
Other: Short term (10 day) low residue diet restriction — Patients will have an unrestricted diet (as opposed to a low residue diet restriction) 10 days after surgery.
  Arms: 10 day low residue diet restriction after surgery
Other: 6 week low residue diet restriction — Patients will be restricted to a low residue diet for 6 weeks after surgery. After this period, their diet will be unrestricted.
  Arms: 6 week low residue diet restriction after surgery

SUMMARY:
The goal of this clinical trial is to learn if a 10 day low-residue diet restriction is better for bowel function and quality of life without increasing complications compared to a 6 week low-residue diet restriction after elective colon resection surgery. The main questions it aims to answer are:

Does a shorter time period of low residue restriction result in a faster return to normal bowel function? Are there any differences in complication rate between a 10 day low-residue diet restriction compared to a 6 week low-residue diet restriction?

Participants will be randomized to one of the two diet plans and will be asked to answer surveys about their bowel function and health care related quality of life at various time points for up to 3 months.

DETAILED DESCRIPTION:
Patients who undergo colon resection surgery are often instructed to adhere to a low residue (low insoluble fiber) diet for at least the first 1-2 weeks after surgery. This approach is based on limited previous literature that associates stool burden in the first three to seven days and the risk of leakage from the new connection in the colon (anastomotic leakage). However, there is no clear consensus on how long this low residue diet should last, and low residue diets can negatively affect bowel function-related quality of life. The investigators hypothesize that resuming an unrestricted diet at an earlier time point (10 days) after surgery will improve bowel function-related quality of life without increasing the risk of leakage or other complications compared to a longer time point (6 weeks). Both time points are within the scope of practice, but many surgeons opt for the longer time point. To answer our hypothesis, the investigators plan to use validated survey instruments pre- and postoperatively (at within 2 weeks preoperatively then 1 week, 3 week, 6 week, and 3 months after the surgery) to assess patient's bowel function and health care-related quality of life. Patients will be consented preoperatively and randomized after their surgeries, no later than the day of discharge from the hospital. The participants will take a survey before surgery then have their surgery as the participants normally would. The participants will also have their post-surgery hospital care as normal and before discharge will be instructed on which diet plan the participants must follow (either 10 days or 6 weeks of low residue diet). Patients who have postoperative issues while in the hospital will be excluded, as the participants usually have different postoperative diet recommendations outside of the typical post-surgical pathway. Other than the surveys and different diet instructions, nothing else will change about their post-surgical care. The results of the surveys for each group will be evaluated in several ways. Summary statistics will be obtained to characterize both the intervention and control group. In addition, the pre and post-surgical results will be compared. Other information will be collected, such as demographic information and complication rate, that will be used to compare both groups as well. These results and the subsequent analysis will address our hypothesis and allow us to either recommend a 10-day period of low residue diet or confirm that the 6-week period is safer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have elective colon resection with anastomosis

Exclusion Criteria:

* Patients who have an ostomy as part of their surgery
* Patients who undergo emergency surgery
* Patients who do not follow the enhanced recovery protocol (the standard postoperative protocol for patients undergoing elective colon resection)
* Patients less than 18 years of age
* Vulnerable populations: fetuses, pregnant women, children, cognitively impaired, hospital employees, students, healthy controls, prisoners, and other institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Return to baseline bowel function (Postoperative Low Anterior Resection Syndrome Score - Preoperative Low Anterior Resection Syndrome Score <=5) | Preoperative to 3 months postoperative
  Return to baseline bowel function is defined by comparing the preoperative LARS score (range 0-42) to postoperative LARS score (range 0-42). Return to baseline is defined as a difference equal to or less than 5 when subtracting the postoperative score by the preoperative score.

SECONDARY OUTCOMES:
Bowel Function Related Quality of Life | preoperative to 3 months postoperative
  This is a single question survey asking patients about the impact their bowel function has on their quality of life. These answers will be accumulated and compared across both groups. From better to worse, the answers are: A) not at all, B) very little, C) somewhat, D) a lot.
Health Care Related Quality of Life | preoperative to 3 months postoperative
  This outcome measure is based on 36-Item Short Form Survey Instrument (SF-36) scores which will be averaged, separated in its components, and compared across groups. Each component is scored from 0 - 100 based on responses from the participants, with 100 being the best possible score.

OTHER OUTCOMES:
Complication Rate | Preoperative to 2 years postoperative
  Complications, if any occur, will be recorded for each group and incidence of complications will be compared across groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Zimmern, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Hospital, New Hyde Park, New York

IPD SHARING:
Plan to Share IPD: No
We do not intend to share IPD with other researchers. Data deidentified through REDCap may be shared upon publication of results if requested by the journal and in compliance with IRB requirements.

REFERENCES:
- [Background] Kawada K, Wada T, Yamamoto T, Itatani Y, Hida K, Obama K. Correlation between Colon Perfusion and Postoperative Fecal Output through a Transanal Drainage Tube during Laparoscopic Low Anterior Resection. Cancers (Basel). 2022 May 8;14(9):2328. doi: 10.3390/cancers14092328. PMID 35565456
- [Background] Lau C, Phillips E, Bresee C, Fleshner P. Early use of low residue diet is superior to clear liquid diet after elective colorectal surgery: a randomized controlled trial. Ann Surg. 2014 Oct;260(4):641-7; discussion 647-9. doi: 10.1097/SLA.0000000000000929. PMID 25203881
- [Background] Vanhauwaert E, Matthys C, Verdonck L, De Preter V. Low-residue and low-fiber diets in gastrointestinal disease management. Adv Nutr. 2015 Nov 13;6(6):820-7. doi: 10.3945/an.115.009688. Print 2015 Nov. PMID 26567203
- [Background] Blomquist P, Jiborn H, Zederfeldt B. The effect of relative bowel rest on healing of colonic anastomoses. Breaking strength and collagen in the colonic wall following left colon resection and anastomosis in the rat. Acta Chir Scand. 1984;150(8):671-5. PMID 6532041
- [Background] Uden P, Blomquist P, Jiborn H, Zederfeldt B. Influence of long-term relative bowel rest on the healing of a left colon anastomosis. Dis Colon Rectum. 1988 Nov;31(11):886-91. doi: 10.1007/BF02554855. PMID 3180961
- [Background] Emmertsen KJ, Laurberg S. Low anterior resection syndrome score: development and validation of a symptom-based scoring system for bowel dysfunction after low anterior resection for rectal cancer. Ann Surg. 2012 May;255(5):922-8. doi: 10.1097/SLA.0b013e31824f1c21. PMID 22504191
- [Background] He S, Zhang J, Wang R, Li L, Sun W, Wang J, Deng Y, Liang W, Dou R. Long-term Changes in Low Anterior Resection Syndrome in Survivors of Rectal Cancer: Longitudinal Follow-up of a Randomized Controlled Trial. Dis Colon Rectum. 2024 Jun 1;67(6):834-840. doi: 10.1097/DCR.0000000000003262. Epub 2024 Mar 1. PMID 38426539
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] Wang A, Robitaille S, Liberman S, Feldman LS, Fiore JF Jr, Lee L. Does the Low Anterior Resection Syndrome Score Accurately Represent the Impact of Bowel Dysfunction on Health-Related Quality of Life? J Gastrointest Surg. 2023 Jan;27(1):114-121. doi: 10.1007/s11605-022-05481-z. Epub 2022 Oct 17. PMID 36253504
- [Background] Battersby NJ, Juul T, Christensen P, Janjua AZ, Branagan G, Emmertsen KJ, Norton C, Hughes R, Laurberg S, Moran BJ; United Kingdom Low Anterior Resection Syndrome Study Group. Predicting the Risk of Bowel-Related Quality-of-Life Impairment After Restorative Resection for Rectal Cancer: A Multicenter Cross-Sectional Study. Dis Colon Rectum. 2016 Apr;59(4):270-80. doi: 10.1097/DCR.0000000000000552. PMID 26953985